CLINICAL TRIAL: NCT07386912
Title: Investigation of the Effects of Oxidized Antigens on the T-Cell Response and the Epigenetic Reprogramming of Neutrophils in Lung Diseases - OXIGENE -
Acronym: OXIGENE
Status: Not yet recruiting | Type: Observational
Sponsor: Research Center Borstel (Other)
Responsible Party: Principal Investigator, Jan Heyckendorf, Prof. Dr. med. Jan Heyckendorf, University Hospital Schleswig-Holstein
Other Study IDs: OXIGENE
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Asthma; COPD; Bacterial Pneumonia; Viral Pneumonia; Tuberculosis
Keywords: neutrophil granulocytes; epigenome; oxidation; antigens
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Pneumonia, Bacterial; Pneumonia, Viral; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Li-heparine plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Asthma: Patients with Asthma
  Interventions: Other: Characterization of the neutrophil granulocyte epigenome
- COPD: Patients with chronic obstructive pulmonary disease
  Interventions: Other: Characterization of the neutrophil granulocyte epigenome
- Viral pneumonia: Patients suffering from viral pneumonia, e.g. COVID-19 or Influenza
  Interventions: Other: Characterization of the neutrophil granulocyte epigenome
- Bacterial pneumonia: Patients suffering from bacterial pneumonia
  Interventions: Other: Characterization of the neutrophil granulocyte epigenome
- Tuberculosis: Patients treated for tuberculosis
  Interventions: Other: Characterization of the neutrophil granulocyte epigenome; Other: Characterization of the T-cell immune response to to various oxidatively modified mycobacterial antigens

INTERVENTIONS:
Other: Characterization of the neutrophil granulocyte epigenome — Characterization of epigenomic differences in neutrophils from patients with different lung diseases (asthma, COPD, pneumonia, tuberculosis, and viral pulmonary infections such as COVID-19 and influenza) by identifying disease-specific epigenetic and functional signatures
Other: Characterization of the T-cell immune response to to various oxidatively modified mycobacterial antigens — Investigation of the response (activation/stimulation) of antigen-specific T cells from patients with tuberculosis to various oxidatively modified mycobacterial antigens, with the aim of determining whether changes in the redox status of these antigens measurably influence the adaptive immune response.
  Groups: Tuberculosis

SUMMARY:
The OXIGENE study is a research project that aims to better understand how the immune system behaves in people with lung diseases such as asthma, COPD, pneumonia, tuberculosis, and viral lung infections. By analyzing a single blood sample, the study examines how certain immune cells react during inflammation and infection, and whether lasting changes in these cells influence how strongly the body responds to disease. Although participants do not receive direct medical benefit, the results may help improve future diagnosis and treatment of lung diseases by providing deeper insight into immune responses.

DETAILED DESCRIPTION:
The OXIGENE study is an observational research project that explores how the human immune system responds in different lung diseases, including asthma, COPD, pneumonia, tuberculosis, and viral lung infections such as COVID-19 or influenza. The study focuses on two key components of the immune system: neutrophils, which are among the first immune cells to respond to inflammation, and T cells, which play an important role in longer-term immune defense. Researchers investigate whether neutrophils show lasting changes in their behavior during lung disease and how these changes may differ depending on the type of illness or individual patient characteristics. In people with tuberculosis, the study also examines whether chemical changes to bacterial proteins caused by inflammation influence how strongly T cells are activated.

Participation in the study involves a single blood draw, similar to a routine blood test, with no medications, interventions, or follow-up visits required. The study does not provide direct medical benefit to participants, but the risks are minimal and limited to those associated with blood sampling. By improving the understanding of how immune responses are altered in lung diseases, the OXIGENE study aims to generate knowledge that could support the development of better diagnostic tools and more targeted treatments for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an acute or chronic inflammatory lung disease, infectious or non-infectious, including asthma, COPD, pneumonia, tuberculosis, or viral pulmonary infection (e.g., COVID-19, influenza).
* Age ≥ 18 years at the time of informed consent.
* Ability to provide informed consent and consent to the collection and processing of clinical and laboratory data, as well as to the analysis of blood samples as part of study participation.
* Sufficient physical condition to undergo a single venous blood draw (approximately 50 mL), as assessed by the treating physician.

Exclusion Criteria:

* Active malignant disease or ongoing cancer therapy (e.g., chemotherapy or immunotherapy), due to potential immunological confounding.
* Immunosuppressive therapy or known severe immunodeficiency that could interfere with the interpretation of cellular immune responses.
* Pregnancy or breastfeeding, for general research-ethical reasons and to protect vulnerable populations.
* Acute unstable clinical condition that, in the opinion of the treating physician, makes study participation unreasonable.
* Known intolerance to blood sampling or relevant hematological disorders that could compromise the safety or feasibility of venipuncture.
* Lack of capacity to provide informed consent or insufficient understanding of the study content despite supportive explanation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes only adult patients (≥18 years) with lung diseases who are capable of providing informed consent and are medically fit for a single venous blood draw. Minors, healthy volunteers, and adults lacking the capacity to consent are not included, as consent by legal representatives is not provided for, and the study involves no interventions beyond blood sampling. Women of childbearing potential may participate regardless of contraceptive use, as study participation poses no additional risk. Patients with insufficient German language proficiency may also be included; in such cases, study information is provided orally in a language the participant fully understands by a qualified translator, with the translation process documented, and written consent is given using the German-language consent form once full understanding has been ensured, allowing all participants to make an informed and voluntary decision.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of the neutrophil granulocyte epigenome | 2030
  Stratification of patients with different lung diseases based on epigenetic signatures of neutrophils: Epigenetics: identification of disease-specific differences in DNA methylation patterns and transcriptional profiles (RNA sequencing).
Characterization of functional signatures | 2030
  Stratification of patients with different lung diseases based on functional signatures of neutrophils:
  Functional reactivity: quantitative assessment of reactive oxygen species production (oxidative burst) and cellular cell death (e.g., Sytox Green, Annexin V/PI) following stimulation with defined stimuli (e.g., PMA, LPS, Gram-positive/Gram-negative bacteria, BCG, Mycobacterium tuberculosis).

SECONDARY OUTCOMES:
Influence of demographic and clinical variables | 2030
  Correlation of demographic and clinical variables (age, sex, disease severity, medication, comorbidities) with epigenetic and functional parameters
Identification of subgroups within diseases | 2030
  Exploratory identification of subgroups with characteristic or divergent profiles within the studied patient cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Jan Heyckendorf, Prof. Dr. med., Principal Investigator — University Hospital Schleswig-Holstein
Locations (2):
- Germany (2):
  - Medical Service Center MVZ, Research Center Borstel, Leibniz Lung Center, Borstel, Schleswig-Holstein
  - Department of Pulmonology, University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared upon reasonable request. Please contact the prinicpal investigator.